CLINICAL TRIAL: NCT04472234
Title: Could the Consumption of Water From Plastic Bottles Affect the Embryo Grade and Clinical Pregnancy Rate Obtained With IVF/ICSI in Unexplained Infertility
Brief Title: BPA Levels Relationship With IVF/ICSI Outcomes in Unexplained Infertility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nefise Nazlı YENIGUL (Other)
Responsible Party: Sponsor-Investigator, Nefise Nazlı YENIGUL, Ph.D. Assistant Professor Department of Obstetrics and Gynecolog, Sanliurfa Mehmet Akif Inan Education and Research Hospital
Organization: Sanliurfa Mehmet Akif Inan Education and Research Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019/15
Record Dates: First submitted 2020-07-01; First posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Infertility Unexplained; IVF; Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BPA level (Other): BPA (Bisfenol A) in urine, blood and follicle fluid samples
  Interventions: Other: BPA levels

INTERVENTIONS:
Other: BPA levels — BPA (Bisfenol A) in urine, blood and follicle fluid samples

SUMMARY:
The relationship between BPA elevation in urine, blood, and follicle fluid and embryo quality, IVF/ICSI outcomes.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 23-33 years who underwent IVF due to unexplained infertility
* patients provided urine, blood, and follicle fluid (FF) samples on the oocyte retrieval day
* patients who did not smoke or use alcohol
* patients did not work in the plastic industry

Exclusion Criteria:

* patients who underwent IVF due to low ovarian reserve or tubal factor or male factor indications
* patients diagnosed with endometriosis
* patients with freeze-all cycles
* women with metabolic disease (such as hypertension or diabetes mellitus)
* patients with a known genetic problem (male or female)

Ages: 23 Years to 33 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Exposure to BPA | 6 month
  Concentrations of Bisphenol A (BPA) will be quantified in the ürine, blood plasma, and follicular fluid (individual and pooled samples) by use of ELİSA test in women with unexplained infertility

CONTACTS AND LOCATIONS:
Locations (1):
- Nefise Nazlı YENIGUL, Sanliurfa, Turkey (Türkiye)